CLINICAL TRIAL: NCT01910402
Title: A Phase IIIb, Randomized, Open-label Study of the Safety and Efficacy of Dolutegravir/Abacavir/Lamivudine Once Daily Compared to Atazanavir and Ritonavir Plus Tenofovir/Emtricitabine Once Daily in HIV-1 Infected Antiretroviral Therapy Naïve Women
Brief Title: A Study to Determine Safety and Efficacy of Dolutegravir/Abacavir/Lamivudine (DTG/ABC/3TC) in Human Immunodeficiency Virus (HIV)-1 Infected Antiretroviral Therapy (ART) Naïve Women (ARIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117172; 2012-005823-34 (EudraCT Number)
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: antiretroviral therapy naïve; women; once daily; HIV infection; atazanavir; tenofovir/emtricitabine; dolutegravir/abacavir/lamivudine fixed dose combination; integrase inhibitor; ritonavir
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir; Atazanavir Sulfate; Ritonavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DTG/ABC/3TC FDC (Experimental): As per the randomization schedule subjects will be administered with DTG/ABC/3TC (50mg/600mg/300mg) FDC tablet OD up to Week 48 and if continued if applicable in the Continuation Phase. DTG/ABC/3TC FDC may be administered with or without food
  Interventions: Drug: Dolutegravir/abacavir/lamivudine FDC
- ATV +RTV +TDF/FTC FDC (Active Comparator): As per the randomization schedule subjects will be administered with ATV (300mg capsule) +RTV (100mg tablet) + TDF/FTC (300mg/200mg tablet) FDC OD up to Week 48. ATV+RTV+ TDF/FTC FDC must be taken with food
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Tenofovir/emtricitabine FDC

INTERVENTIONS:
Drug: Dolutegravir/abacavir/lamivudine FDC — Dolutegravir/abacavir/lamivudine FDC tablets, 50 mg/600 mg/300 mg
  Arms: DTG/ABC/3TC FDC
Drug: Atazanavir — Atazanavir capsule 300 mg
  Arms: ATV +RTV +TDF/FTC FDC
Drug: Ritonavir — Ritonavir tablet 100 mg
  Arms: ATV +RTV +TDF/FTC FDC
Drug: Tenofovir/emtricitabine FDC — Tenofovir/emtricitabine FDC tablet 300 mg/200 mg of FTC
  Arms: ATV +RTV +TDF/FTC FDC

SUMMARY:
This study is designed to demonstrate the non-inferior antiviral activity of DTG/ABC/3TC fixed dose combination (FDC) once daily (OD) compared to atazanavir plus ritonavir (ATV+RTV) and tenofovir disoproxil fumarate/emtricitabine fixed dose combination (TDF/FTC FDC) OD in HIV-1 infected, ART-naïve women over 48 weeks. This study will also characterize the safety and tolerability of DTG/ABC/3TC FDC compared to ATV+RTV+TDF/FTC FDC. Sufficient number of subjects will be screened in order to ensure a total of approximately 474 subjects will be randomized (237 in each study arm)

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected females (gender at birth) >=18 years of age
* Women capable of becoming pregnant must use appropriate contraception during the study (as defined by the protocol)
* HIV-1 infection as documented by Screening plasma HIV-1 RNA >=500 c/mL.
* Documentation that the subject is negative for the HLA-B*5701 allele.
* Antiretroviral-naïve (<=10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection).
* Signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Women who plan to become pregnant during the first 48 weeks of the study
* Any subject who has had a medical intervention for gender reassignment
* Any evidence of an active Centers for Disease Control and Prevention (CDC) Category C disease
* Subjects with any degree of hepatic impairment
* Subjects positive for hepatitis B at Screening, or anticipated need for HCV therapy during the study
* History or presence of allergy to the study drugs or their components or drugs of their class
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia
* poses a significant suicidality risk
* History of osteoporosis with fracture or requiring pharmacologic therapy
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses;
* Treatment with any agent, with documented activity against HIV-1 in vitro within 28 days of first dose of investigational product (IP)
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of IP
* Any evidence of primary viral resistance based on the presence of any major resistance-associated mutation in the Screening result or, if known, any historical resistance test result
* Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 lipid abnormalities (total cholesterol, triglycerides, High Density Lipoprotein (HDL) cholesterol, Low Density Lipoprotein (LDL) cholesterol)
* Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound
* Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN), or ALT ≥ 3xULN and bilirubin ≥ 1.5xULN (with >35% direct bilirubin)
* Subject has CrCL of <50 mL/min via Cockroft-Gault method
* Corrected QT interval (QTc (Bazett)) ≥450msec or QTc (Bazett) ≥480msec for subjects with bundle branch block.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2013-08-22 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (80):
- United States (34):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Lynchburg, Virginia
- Argentina (3):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (3):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Italy (6):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Busto Arsizio (VA), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
- Mexico (2):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, México
- Portugal (3):
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Puerto Rico (3):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, Rio Piedras
  - GSK Investigational Site, San Juan
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Toliyatti
- South Africa (2):
  - GSK Investigational Site, Observatory, Cape Town, Western Province
  - GSK Investigational Site, Mamelodi East
- Spain (9):
  - GSK Investigational Site, (Móstoles) Madrid
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Seville
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Nonthaburi
- United Kingdom (4):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, London
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Tooting, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on ViiV's data sharing criteria can be found at: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/

REFERENCES:
- [Derived] Orrell C, Hagins DP, Belonosova E, Porteiro N, Walmsley S, Falco V, Man CY, Aylott A, Buchanan AM, Wynne B, Vavro C, Aboud M, Smith KY; ARIA study team. Fixed-dose combination dolutegravir, abacavir, and lamivudine versus ritonavir-boosted atazanavir plus tenofovir disoproxil fumarate and emtricitabine in previously untreated women with HIV-1 infection (ARIA): week 48 results from a randomised, open-label, non-inferiority, phase 3b study. Lancet HIV. 2017 Dec;4(12):e536-e546. doi: 10.1016/S2352-3018(17)30095-4. Epub 2017 Jul 17. PMID 28729158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consists of a Screening (14-28 days), Randomized (48 weeks) and Continuation (Cont.) Phase. Participants were said to have completed the study if they completed the Randomized phase and did not enter the Cont. Phase. Participants entering the Cont. Phase were said to have completed the study if they completed both phases of the study.
Pre-assignment Details: A total of 499 participants were randomized to receive dolutegravir(DTG)/abacavir(ABC)/lamivudine(3TC) fixed dose combination(FDC) or combination of atazanavir(ATV), Ritonavir(RTV) and FDC of tenofovir disoproxil fumarate/emtricitabine(TDF/FTC). Two participants from each DTG/ABC/3TC and ATV+RTV+TDF/FTC groups were randomized but not treated. A total of 495 participants received at least single dose of investigational products(IP) and were included in Intent-to-Treat Exposed(ITT-E) Population.
Groups:
- DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase: Participants received fixed dose combination (FDC) of DTG 50 milligram (mg)/ABC 600 mg/3TC 300 mg tablet once daily orally for 48 weeks in the Randomization Phase.
- ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase: Participants received ATV 300 mg capsule, RTV 100 mg tablet, TDF 300 mg/ FTC 200 mg FDC tablet once daily orally for 48 weeks during Randomized Phase.
- DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase: Participants received DTG 50 mg/ABC 600 mg/3TC 300 mg once daily orally in the Continuation Phase until it was either locally approved or commercial supplies were available.
Period: Randomized Phase (Up to 48 Weeks)
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Started (Randomized) | 250 | 249 | 0
ITT-E Population | 248 | 247 | 0
Completed | 206 | 192 | 0
Not Completed | 44 | 57 | 0
Not completed — Adverse Event | 10 | 18 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lack of Efficacy | 5 | 4 | 0
Not completed — Lost to Follow-up | 11 | 13 | 0
Not completed — Withdrawal by Subject | 5 | 7 | 0
Not completed — Randomized, but did not receive treatment | 2 | 2 | 0
Not completed — Protocol Deviation | 10 | 13 | 0
Period: Continuation Phase(From Weeks 48 to 432)
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Started | 0 | 0 | 149 (149 participants from the Randomized Phase entered in the Continuation Phase)
Completed | 0 | 0 | 113
Not Completed | 0 | 0 | 36
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 7
Not completed — Lost to Follow-up | 0 | 0 | 8
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 15

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for members of the ITT-E Population which comprised of all randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase | Total
Number analyzed (Participants) | 248 | 247 | 495
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (11.15) | 37.8 (10.14) | 37.9 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 247 | 495
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 102 | 108 | 210
  American Indian Or Alaskan Native | 6 | 7 | 13
  Asian - Central/South Asian Heritage | 2 | 0 | 2
  Asian - East Asian Heritage | 0 | 1 | 1
  Asian - South East Asian Heritage | 20 | 22 | 42
  Native Hawaiian Or Other Pacific Islander | 1 | 0 | 1
  White - Arabic/North African Heritage | 3 | 3 | 6
  White - White/Caucasian/European Heritage | 112 | 104 | 216
  Mixed Race | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/mL at Week 48
Description: Percentage of participants with plasma human immunodeficiency virus type 1(HIV-1) ribonucleic acid (RNA) <50 copies per milliliter (c/mL) were assessed at Week 48 using the Snapshot algorithm. Analysis was performed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for Baseline plasma HIV-1 RNA ( =<vs. >100,000 c/mL) and CD4+ cell count (=<350 cells per millimeter cube (cells/mm^3) or >350 cells/mm^3). Intent-to-Treat Exposed (ITT-E) Population comprised of all randomized participants who received at least one dose of study medication. Percentage values are rounded off.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Percentage of participants | 82 | 71
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Non-Inferiority or Equivalence — Hypothesis was to show that the antiviral effect of the DTG/ABC/3TC FDC administered QD was non-inferior to QD ATV+RTV+TDF/FTC FDC. Non-inferiority was concluded if the lower bound of a two-sided 95% confidence interval for the difference in response rates between the two treatment arms was greater than -12%; p = 0.005, Cochran-Mantel-Haenszel — If the primary and PP analyses both demonstrated non-inferiority, then as per pre-specified analysis, superiority of DTG/ABC/3TC FDC versus ATV+RTV+TDF/FTC FDC was tested in the ITT-E population at the 2-sided 5% level of significance; Adjusted difference in proportion = 10.5, 95% CI 2-sided [3.1 to 17.8]

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 and <400 c/mL Over Time-Randomized Phase
Description: Percentage of participants with plasma HIV-1 RNA <50 and <400 c/mL were assessed at Baseline, Weeks 4, 12, 24 , 36 and 48 using the Snapshot algorithm (Missing, Switch or Discontinuation = Failure). The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Percentage values are rounded off.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Percentage of participants
  HIV-1 RNA <50 c/mL, Baseline (Day 1) | 0 | 0
  HIV-1 RNA <50 c/mL, Week 4 | 64 | 13
  HIV-1 RNA <50 c/mL, Week 12 | 81 | 49
  HIV-1 RNA <50 c/mL, Week 24 | 85 | 77
  HIV-1 RNA <50 c/mL, Week 36 | 85 | 77
  HIV-1 RNA <50 c/mL, Week 48 | 82 | 71
  HIV-1 RNA <400 c/mL, Baseline (Day 1) | 1 | 1
  HIV-1 RNA <400 c/mL, Week 4 | 90 | 54
  HIV-1 RNA <400 c/mL, Week 12 | 91 | 84
  HIV-1 RNA <400 c/mL, Week 24 | 88 | 82
  HIV-1 RNA <400 c/mL, Week 36 | 86 | 81
  HIV-1 RNA <400 c/mL, Week 48 | 83 | 76

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL in Continuation Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Percentage of participants with plasma HIV-1 RNA <50 c/mL were reported. Percentage values are rounded off.
Time Frame: Week 96 and Week 432
Population: ITT-E Population. Only those participants with data available at indicated time points were analyzed (represented by n=X in category titles)
Measure: Number; unit: Percentage of participants
Groups:
- DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase: Participants received DTG 50 mg/ABC 600 mg/3TC 300 mg QD in the Continuation Phase until it was either locally approved or commercial supplies were available.
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Percentage of participants
  Week 96, n=99: number analyzed (Participants) | 99
  Week 96, n=99 | 100
  Week 432, n=3: number analyzed (Participants) | 3
  Week 432, n=3 | 100

4. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA at Indicated Time Points-Randomized Phase
Description: Change from the Baseline in plasma HIV-1 RNA were assessed at indicated time points. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Log10 copies/mL
  Week 4, n=245, 238: number analyzed (Participants) | 245 | 238
  Week 4, n=245, 238 | -2.591 (0.8015) | -1.923 (0.5330)
  Week 12, n=236, 226: number analyzed (Participants) | 236 | 226
  Week 12, n=236, 226 | -2.756 (0.8920) | -2.541 (0.7373)
  Week 24, n=225, 212: number analyzed (Participants) | 225 | 212
  Week 24, n=225, 212 | -2.789 (0.9160) | -2.726 (0.8890)
  Week 36, n=221, 204: number analyzed (Participants) | 221 | 204
  Week 36, n=221, 204 | -2.838 (0.8589) | -2.772 (0.8451)
  Week 48, n=207, 192: number analyzed (Participants) | 207 | 192
  Week 48, n=207, 192 | -2.874 (0.8035) | -2.752 (0.8433)

5. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA at Indicated Time Points-Continuation Phase
Description: as for outcome 4
Time Frame: Baseline (Day 1), Week 96 and Week 432
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Log10 copies/mL
  Week 96, n=99: number analyzed (Participants) | 99
  Week 96, n=99 | -2.911 (0.7970)
  Week 432, n=3: number analyzed (Participants) | 3
  Week 432, n=3 | -3.107 (0.7659)

6. Secondary Outcome: Absolute Values in Plasma HIV-1 RNA at Indicated Time Points-Randomized Phase
Description: Absolute Values in plasma HIV-1 RNA were assessed at indicated time points. The Baseline value was defined as the latest pre-dose assessment (Day 1) value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Log10 copies/mL
  Baseline (Day 1), n=248, 247 | 4.481 (0.8111) | 4.441 (0.8023)
  Week 4, n=245, 238: number analyzed (Participants) | 245 | 238
  Week 4, n=245, 238 | 1.895 (0.6872) | 2.516 (0.6193)
  Week 12, n=236, 226: number analyzed (Participants) | 236 | 226
  Week 12, n=236, 226 | 1.748 (0.5458) | 1.908 (0.4926)
  Week 24, n=225, 212: number analyzed (Participants) | 225 | 212
  Week 24, n=225, 212 | 1.724 (0.5935) | 1.710 (0.4484)
  Week 36, n=221, 204: number analyzed (Participants) | 221 | 204
  Week 36, n=221, 204 | 1.666 (0.3982) | 1.658 (0.3362)
  Week 48, n=207, 192: number analyzed (Participants) | 207 | 192
  Week 48, n=207, 192 | 1.619 (0.1986) | 1.657 (0.2743)

7. Secondary Outcome: Absolute Values in Plasma HIV-1 RNA at Indicated Time Points-Continuation Phase
Description: Absolute Values in plasma HIV-1 RNA were assessed at indicated time points.
Time Frame: Week 96 and Week 432
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Log10 copies/mL
  Week 96, n=99: number analyzed (Participants) | 99
  Week 96, n=99 | 1.591 (0.0080)
  Week 432, n=3: number analyzed (Participants) | 3
  Week 432, n=3 | 1.590 (0.0000)

8. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Indicated Timepoints-Randomized Phase
Description: Change from Baseline in cluster of differentiation 4 (CD4+) cell count were assessed at indicated time points. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Cells per cubic millimeter
  Week 4, n=245, 237: number analyzed (Participants) | 245 | 237
  Week 4, n=245, 237 | 94.9 (140.02) | 73.7 (108.15)
  Week 12, n=236, 224: number analyzed (Participants) | 236 | 224
  Week 12, n=236, 224 | 143.8 (142.19) | 124.4 (133.60)
  Week 24, n=226, 210: number analyzed (Participants) | 226 | 210
  Week 24, n=226, 210 | 200.6 (162.37) | 163.0 (126.67)
  Week 36, n=219, 204: number analyzed (Participants) | 219 | 204
  Week 36, n=219, 204 | 230.7 (163.61) | 191.4 (167.24)
  Week 48, n=208, 191: number analyzed (Participants) | 208 | 191
  Week 48, n=208, 191 | 248.8 (172.01) | 230.7 (189.59)

9. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Indicated Timepoints-Continuation Phase
Description: Change from Baseline in cluster of differentiation 4(CD4+) cell count were assessed at indicated time points. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 96, Week 432
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Cells per cubic millimeter
  Week 96, n=99: number analyzed (Participants) | 99
  Week 96, n=99 | 286.5 (196.77)
  Week 432, n=3: number analyzed (Participants) | 3
  Week 432, n=3 | 254.7 (342.31)

10. Secondary Outcome: Absolute Values in CD4+ Cell Count at Indicated Timepoints-Randomized Phase
Description: Absolute values in CD4+ cell count were assessed at indicated time points. The Baseline value was defined as the latest pre-dose assessment (Day 1) value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Cells per cubic millimeter
  Baseline (Day 1), n=248, 247 | 369.7 (225.67) | 380.3 (223.60)
  Week 4, n=245, 237: number analyzed (Participants) | 245 | 237
  Week 4, n=245, 237 | 465.0 (252.51) | 455.1 (244.62)
  Week 12, n=236, 224: number analyzed (Participants) | 236 | 224
  Week 12, n=236, 224 | 509.5 (276.79) | 506.2 (266.84)
  Week 24, n=226, 210: number analyzed (Participants) | 226 | 210
  Week 24, n=226, 210 | 563.8 (303.10) | 542.5 (265.69)
  Week 36, n=219, 204: number analyzed (Participants) | 219 | 204
  Week 36, n=219, 204 | 592.8 (291.62) | 569.2 (299.77)
  Week 48, n=208, 191: number analyzed (Participants) | 208 | 191
  Week 48, n=208, 191 | 608.8 (298.95) | 608.5 (302.58)

11. Secondary Outcome: Absolute Values in CD4+ Cell Count at Indicated Timepoints-Continuation Phase
Description: Absolute values in CD4+ cell count were assessed at indicated time points.
Time Frame: Week 96 and Week 432
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Cells per cubic millimeter
  Week 96, n=99: number analyzed (Participants) | 99
  Week 96, n=99 | 635.3 (285.85)
  Week 432, n=3: number analyzed (Participants) | 3
  Week 432, n=3 | 553.0 (341.63)

12. Secondary Outcome: Change From Baseline in Carbon Dioxide, Electrolytes, Lipids, Glucose, Urea at Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (Day 1), Weeks 4, 12, 24, 36 and 48. Change from Baseline in carbon dioxide, electrolytes (chloride, hyperkalemia, hypernatremia, hypokalemia, hyponatremia, phosphate, potassium, sodium), lipids (cholesterol [CHLS], high density lipoprotein [HDL] CHLS direct, low density lipoprotein (LDL) CHLS calculation, LDL CHLS direct, triglycerides), glucose (hyperglycaemia, hypoglycaemia) and urea are summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value. Laboratory parameters were assessed in Safety Population which comprised of all participants who received at least one dose of study treatment.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Millimoles per liter
  Carbon Dioxide, Week 4, n= 244, 237: number analyzed (Participants) | 244 | 237
  Carbon Dioxide, Week 4, n= 244, 237 | -0.4 (2.29) | 0.6 (2.2)
  Carbon Dioxide, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Carbon Dioxide, Week 12, n= 236, 226 | -0.2 (2.2) | 0.8 (2.19)
  Carbon Dioxide, Week 24, n= 224, 212: number analyzed (Participants) | 224 | 212
  Carbon Dioxide, Week 24, n= 224, 212 | -0.5 (2.31) | 0.3 (2.38)
  Carbon Dioxide, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Carbon Dioxide, Week 36, n= 219, 204 | 0 (2.34) | 0.6 (2.5)
  Carbon Dioxide, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Carbon Dioxide, Week 48, n= 208, 192 | -0.6 (2.55) | 0.4 (2.46)
  Chloride, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Chloride, Week 4, n= 245, 237 | 0.6 (2.42) | -0.5 (2.68)
  Chloride, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Chloride, Week 12, n= 236, 226 | 1 (2.51) | 0.2 (2.58)
  Chloride, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Chloride, Week 24, n= 225, 212 | 0.7 (2.71) | -0.1 (2.58)
  Chloride, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Chloride, Week 36, n= 219, 204 | 0.9 (2.65) | 0 (2.96)
  Chloride, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Chloride, Week 48, n= 208, 192 | 0.7 (2.42) | 0 (2.63)
  CHLS, Week 4, n= 1, 3: number analyzed (Participants) | 1 | 3
  CHLS, Week 4, n= 1, 3 | -0.1 (NA) — NA indicates standard deviation could not be calculated for a single participant | -0.017 (0.446)
  CHLS, Week 12, n= 224, 221: number analyzed (Participants) | 224 | 221
  CHLS, Week 12, n= 224, 221 | 0.298 (0.7492) | -0.058 (0.7137)
  CHLS, Week 24, n= 218, 201: number analyzed (Participants) | 218 | 201
  CHLS, Week 24, n= 218, 201 | 0.317 (0.7254) | -0.001 (0.7456)
  CHLS, Week 36, n= 205, 191: number analyzed (Participants) | 205 | 191
  CHLS, Week 36, n= 205, 191 | 0.33 (0.7328) | 0 (0.7509)
  CHLS, Week 48, n= 195, 175: number analyzed (Participants) | 195 | 175
  CHLS, Week 48, n= 195, 175 | 0.447 (0.7441) | 0.109 (0.7647)
  Glucose, Week 12, n= 226, 224: number analyzed (Participants) | 226 | 224
  Glucose, Week 12, n= 226, 224 | 0.3 (1.359) | 0.22 (1.234)
  Glucose, Week 24, n= 219, 204: number analyzed (Participants) | 219 | 204
  Glucose, Week 24, n= 219, 204 | 0.17 (0.811) | 0.26 (1.248)
  Glucose, Week 36, n= 211, 196: number analyzed (Participants) | 211 | 196
  Glucose, Week 36, n= 211, 196 | 0.17 (1.24) | 0.34 (1.753)
  Glucose, Week 48, n= 197, 180: number analyzed (Participants) | 197 | 180
  Glucose, Week 48, n= 197, 180 | 0.18 (1.01) | 0.24 (1.377)
  HDL CHLS, Direct, Week 4, n= 1, 3: number analyzed (Participants) | 1 | 3
  HDL CHLS, Direct, Week 4, n= 1, 3 | -0.1 (NA) — NA indicates standard deviation could not be calculated for a single participant | 0 (0.0529)
  HDL CHLS, Direct, Week 12, n= 224, 221: number analyzed (Participants) | 224 | 221
  HDL CHLS, Direct, Week 12, n= 224, 221 | 0.182 (0.3407) | 0.005 (0.2316)
  HDL CHLS, Direct, Week 24, n= 218, 201: number analyzed (Participants) | 218 | 201
  HDL CHLS, Direct, Week 24, n= 218, 201 | 0.201 (0.2962) | 0.053 (0.2819)
  HDL CHLS, Direct, Week 36, n= 205, 191: number analyzed (Participants) | 205 | 191
  HDL CHLS, Direct, Week 36, n= 205, 191 | 0.204 (0.2943) | 0.036 (0.2848)
  HDL CHLS, Direct, Week 48, n= 195, 175: number analyzed (Participants) | 195 | 175
  HDL CHLS, Direct, Week 48, n= 195, 175 | 0.231 (0.2911) | 0.081 (0.2964)
  Hyperglycaemia, Week 12, n= 226, 224: number analyzed (Participants) | 226 | 224
  Hyperglycaemia, Week 12, n= 226, 224 | 0.3 (1.359) | 0.22 (1.234)
  Hyperglycaemia, Week 24, n= 219, 204: number analyzed (Participants) | 219 | 204
  Hyperglycaemia, Week 24, n= 219, 204 | 0.17 (0.811) | 0.26 (1.248)
  Hyperglycaemia, Week 36, n= 211, 196: number analyzed (Participants) | 211 | 196
  Hyperglycaemia, Week 36, n= 211, 196 | 0.17 (1.24) | 0.34 (1.753)
  Hyperglycaemia, Week 48, n= 197, 180: number analyzed (Participants) | 197 | 180
  Hyperglycaemia, Week 48, n= 197, 180 | 0.18 (1.01) | 0.24 (1.377)
  Hyperkalemia, Week 4, n= 244, 237: number analyzed (Participants) | 244 | 237
  Hyperkalemia, Week 4, n= 244, 237 | -0.01 (0.344) | 0.12 (0.367)
  Hyperkalemia, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Hyperkalemia, Week 12, n= 236, 226 | 0.03 (0.355) | 0.1 (0.39)
  Hyperkalemia, Week 24, n= 224, 212: number analyzed (Participants) | 224 | 212
  Hyperkalemia, Week 24, n= 224, 212 | -0.04 (0.339) | 0.06 (0.372)
  Hyperkalemia, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Hyperkalemia, Week 36, n= 219, 204 | 0.03 (0.332) | 0.13 (0.387)
  Hyperkalemia, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Hyperkalemia, Week 48, n= 208, 192 | -0.04 (0.346) | 0.04 (0.372)
  Hypernatremia, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Hypernatremia, Week 4, n= 245, 237 | 0 (2.11) | -0.5 (2.4)
  Hypernatremia, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Hypernatremia, Week 12, n= 236, 226 | 0.7 (2.3) | 0.1 (2.51)
  Hypernatremia, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Hypernatremia, Week 24, n= 225, 212 | 0.6 (2.3) | 0.2 (2.11)
  Hypernatremia, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Hypernatremia, Week 36, n= 219, 204 | 0.9 (2.32) | 0.2 (2.5)
  Hypernatremia, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Hypernatremia, Week 48, n= 208, 192 | 0.6 (2.24) | 0.5 (2.39)
  Hypoglycaemia, Week 12, n= 226, 224: number analyzed (Participants) | 226 | 224
  Hypoglycaemia, Week 12, n= 226, 224 | 0.3 (1.359) | 0.22 (1.234)
  Hypoglycaemia, Week 24, n= 219, 204: number analyzed (Participants) | 219 | 204
  Hypoglycaemia, Week 24, n= 219, 204 | 0.17 (0.811) | 0.26 (1.248)
  Hypoglycaemia, Week 36, n= 211, 196: number analyzed (Participants) | 211 | 196
  Hypoglycaemia, Week 36, n= 211, 196 | 0.17 (1.24) | 0.34 (1.753)
  Hypoglycaemia, Week 48, n= 197, 180: number analyzed (Participants) | 197 | 180
  Hypoglycaemia, Week 48, n= 197, 180 | 0.18 (1.01) | 0.24 (1.377)
  Hypokalemia, Week 4, n= 244, 237: number analyzed (Participants) | 244 | 237
  Hypokalemia, Week 4, n= 244, 237 | -0.01 (0.344) | 0.12 (0.367)
  Hypokalemia, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Hypokalemia, Week 12, n= 236, 226 | 0.03 (0.355) | 0.1 (0.39)
  Hypokalemia, Week 24, n= 224, 212: number analyzed (Participants) | 224 | 212
  Hypokalemia, Week 24, n= 224, 212 | -0.04 (0.339) | 0.06 (0.372)
  Hypokalemia, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Hypokalemia, Week 36, n= 219, 204 | 0.03 (0.332) | 0.13 (0.387)
  Hypokalemia, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Hypokalemia, Week 48, n= 208, 192 | -0.04 (0.346) | 0.04 (0.372)
  Hyponatremia, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Hyponatremia, Week 4, n= 245, 237 | 0 (2.11) | -0.5 (2.4)
  Hyponatremia, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Hyponatremia, Week 12, n= 236, 226 | 0.7 (2.3) | 0.1 (2.51)
  Hyponatremia, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Hyponatremia, Week 24, n= 225, 212 | 0.6 (2.3) | 0.2 (2.11)
  Hyponatremia, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Hyponatremia, Week 36, n= 219, 204 | 0.9 (2.32) | 0.2 (2.5)
  Hyponatremia, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Hyponatremia, Week 48, n= 208, 192 | 0.6 (2.24) | 0.5 (2.39)
  LDL CHLS Calculation, Week 4, n= 1, 3: number analyzed (Participants) | 1 | 3
  LDL CHLS Calculation, Week 4, n= 1, 3 | 0.08 (NA) — NA indicates standard deviation could not be calculated for a single participant | -0.123 (0.5255)
  LDL CHLS Calculation, Week 12, n= 221, 219: number analyzed (Participants) | 221 | 219
  LDL CHLS Calculation, Week 12, n= 221, 219 | 0.125 (0.6045) | -0.14 (0.6114)
  LDL CHLS Calculation, Week 24, n= 213, 201: number analyzed (Participants) | 213 | 201
  LDL CHLS Calculation, Week 24, n= 213, 201 | 0.111 (0.6209) | -0.111 (0.6188)
  LDL CHLS Calculation, Week 36, n= 201, 188: number analyzed (Participants) | 201 | 188
  LDL CHLS Calculation, Week 36, n= 201, 188 | 0.112 (0.6385) | -0.099 (0.6049)
  LDL CHLS Calculation, Week 48, n= 190, 175: number analyzed (Participants) | 190 | 175
  LDL CHLS Calculation, Week 48, n= 190, 175 | 0.213 (0.6499) | -0.021 (0.6227)
  LDL CHLS, Direct, Week 12, n= 0, 1: number analyzed (Participants) | 0 | 1
  LDL CHLS, Direct, Week 12, n= 0, 1 |  | -0.44 (NA) — NA indicates standard deviation could not be calculated for a single participant
  LDL CHLS, Direct, Week 24, n= 1, 0: number analyzed (Participants) | 1 | 0
  LDL CHLS, Direct, Week 24, n= 1, 0 | -0.64 (NA) — NA indicates standard deviation could not be calculated for a single participant |
  LDL CHLS, Direct, Week 36, n= 1, 0: number analyzed (Participants) | 1 | 0
  LDL CHLS, Direct, Week 36, n= 1, 0 | -0.23 (NA) — NA indicates standard deviation could not be calculated for a single participant |
  LDL CHLS, Direct, Week 48, n= 0, 0: number analyzed (Participants) | 0 | 0
  Phosphate, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Phosphate, Week 4, n= 245, 237 | 0 (0.1461) | -0.032 (0.1726)
  Phosphate, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Phosphate, Week 12, n= 236, 226 | 0.02 (0.1694) | 0.026 (0.1634)
  Phosphate, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Phosphate, Week 24, n= 225, 212 | 0.021 (0.1628) | 0.026 (0.1701)
  Phosphate, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Phosphate, Week 36, n= 219, 204 | 0.029 (0.1736) | 0.009 (0.1675)
  Phosphate, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Phosphate, Week 48, n= 208, 192 | 0.016 (0.1736) | 0 (0.1673)
  Potassium, Week 4, n= 244, 237: number analyzed (Participants) | 244 | 237
  Potassium, Week 4, n= 244, 237 | -0.01 (0.344) | 0.12 (0.367)
  Potassium, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Potassium, Week 12, n= 236, 226 | 0.03 (0.355) | 0.1 (0.39)
  Potassium, Week 24, n= 224, 212: number analyzed (Participants) | 224 | 212
  Potassium, Week 24, n= 224, 212 | -0.04 (0.339) | 0.06 (0.372)
  Potassium, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Potassium, Week 36, n= 219, 204 | 0.03 (0.332) | 0.13 (0.387)
  Potassium, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Potassium, Week 48, n= 208, 192 | -0.04 (0.346) | 0.04 (0.372)
  Sodium, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Sodium, Week 4, n= 245, 237 | 0 (2.11) | -0.5 (2.4)
  Sodium, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Sodium, Week 12, n= 236, 226 | 0.7 (2.3) | 0.1 (2.51)
  Sodium, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Sodium, Week 24, n= 225, 212 | 0.6 (2.3) | 0.2 (2.11)
  Sodium, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Sodium, Week 36, n= 219, 204 | 0.9 (2.32) | 0.2 (2.5)
  Sodium, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Sodium, Week 48, n= 208, 192 | 0.6 (2.24) | 0.5 (2.39)
  Triglycerides, Week 4, n= 1, 3: number analyzed (Participants) | 1 | 3
  Triglycerides, Week 4, n= 1, 3 | -0.18 (NA) — NA indicates standard deviation could not be calculated for a single participant | 0.237 (0.2491)
  Triglycerides, Week 12, n= 224, 221: number analyzed (Participants) | 224 | 221
  Triglycerides, Week 12, n= 224, 221 | -0.04 (0.6861) | 0.167 (0.7074)
  Triglycerides, Week 24, n= 218, 201: number analyzed (Participants) | 218 | 201
  Triglycerides, Week 24, n= 218, 201 | 0.036 (0.7108) | 0.125 (0.6132)
  Triglycerides, Week 36, n= 205, 191: number analyzed (Participants) | 205 | 191
  Triglycerides, Week 36, n= 205, 191 | 0.037 (0.6732) | 0.157 (0.6785)
  Triglycerides, Week 48, n= 195, 175: number analyzed (Participants) | 195 | 175
  Triglycerides, Week 48, n= 195, 175 | 0.018 (0.8158) | 0.107 (0.5527)
  Urea, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Urea, Week 4, n= 245, 237 | -0.04 (1.085) | 0.1 (1.313)
  Urea, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Urea, Week 12, n= 236, 226 | 0.08 (1.097) | 0.16 (1.409)
  Urea, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Urea, Week 24, n= 225, 212 | 0.03 (1.187) | 0.12 (1.283)
  Urea, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Urea, Week 36, n= 219, 204 | 0.08 (1.236) | -0.03 (1.256)
  Urea, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Urea, Week 48, n= 208, 192 | 0.1 (1.162) | 0.02 (1.179)

13. Secondary Outcome: Change From Baseline in Bilirubin and Creatinine at Indicated Timepoints
Description: Clinical chemistry parameters were assessed at Baseline (Day 1), Weeks 4, 12, 24, 36 and 48. Change from Baseline in bilirubin and creatinine are summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Micromoles per liter
  Bilirubin, Week 4, n= 244, 237: number analyzed (Participants) | 244 | 237
  Bilirubin, Week 4, n= 244, 237 | -0.8 (2.59) | 27.2 (23.15)
  Bilirubin, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Bilirubin, Week 12, n= 236, 226 | -0.6 (2.65) | 22.8 (16.49)
  Bilirubin, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Bilirubin, Week 24, n= 225, 212 | -0.2 (3.06) | 25 (18.38)
  Bilirubin, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Bilirubin, Week 36, n= 219, 204 | -0.2 (3.01) | 23.8 (16.31)
  Bilirubin, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Bilirubin, Week 48, n= 208, 192 | -0.3 (3.08) | 23.7 (17)
  Creatinine, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Creatinine, Week 4, n= 245, 237 | 8.4 (7.057) | 4.89 (7.109)
  Creatinine, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Creatinine, Week 12, n= 236, 226 | 9.2 (8.288) | 5.83 (8.357)
  Creatinine, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Creatinine, Week 24, n= 225, 212 | 9.16 (9.983) | 5.8 (8.063)
  Creatinine, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Creatinine, Week 36, n= 219, 204 | 10.08 (10.473) | 5.37 (9.013)
  Creatinine, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Creatinine, Week 48, n= 208, 192 | 9.29 (8.614) | 5.86 (10.252)

14. Secondary Outcome: Change From Baseline in Albumin at Indicated Timepoints
Description: Clinical chemistry parameters were assessed at Baseline (Day 1), Week 4, 12, 24, 36 and Week 48. Change from Baseline in albumin is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Grams per liter
  Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Week 4, n= 245, 237 | 0.1 (2.36) | -0.5 (2.59)
  Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Week 12, n= 236, 226 | 0.5 (2.95) | 0.1 (2.59)
  Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Week 24, n= 225, 212 | 1.4 (3.2) | 0.8 (2.95)
  Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Week 36, n= 219, 204 | 1.4 (3.09) | 0.6 (2.96)
  Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Week 48, n= 208, 192 | 1.7 (3.17) | 1.3 (3.04)

15. Secondary Outcome: Change From Baseline in Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Creatine Kinase at Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (Day 1), Week 4, 12, 24, 36 and Week 48. Change from Baseline in alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, creatine kinase is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: Safety Population.Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
International units per liter
  Alanine aminotransferase, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Alanine aminotransferase, Week 4, n= 245, 237 | -3.3 (27.54) | -3.4 (15.86)
  Alanine aminotransferase, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Alanine aminotransferase, Week 12, n= 236, 226 | -5.2 (27.51) | -2.3 (20.26)
  Alanine aminotransferase, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Alanine aminotransferase, Week 24, n= 225, 212 | -5.4 (27.92) | -3.7 (20.7)
  Alanine aminotransferase, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Alanine aminotransferase, Week 36, n= 219, 204 | -4.9 (36.11) | -5.3 (20.08)
  Alanine aminotransferase, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Alanine aminotransferase, Week 48, n= 208, 192 | -5.7 (28.54) | -1.5 (31.53)
  Alkaline phosphatase, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Alkaline phosphatase, Week 4, n= 245, 237 | -1.5 (14.56) | 9.4 (28.69)
  Alkaline phosphatase, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Alkaline phosphatase, Week 12, n= 236, 226 | -2.1 (17.1) | 15.1 (30.82)
  Alkaline phosphatase, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Alkaline phosphatase, Week 24, n= 225, 212 | 0.5 (17.86) | 22.4 (41.59)
  Alkaline phosphatase, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Alkaline phosphatase, Week 36, n= 219, 204 | 0.6 (19.19) | 20.4 (30.7)
  Alkaline phosphatase, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Alkaline phosphatase, Week 48, n= 208, 192 | 2.9 (28.05) | 21.9 (25.35)
  Aspartate aminotransferase, Week 4, n= 244, 237: number analyzed (Participants) | 244 | 237
  Aspartate aminotransferase, Week 4, n= 244, 237 | -3.3 (29.8) | -3.6 (18.83)
  Aspartate aminotransferase, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Aspartate aminotransferase, Week 12, n= 236, 226 | -6.2 (21.11) | -4 (13.79)
  Aspartate aminotransferase, Week 24, n= 224, 212: number analyzed (Participants) | 224 | 212
  Aspartate aminotransferase, Week 24, n= 224, 212 | -6.3 (22.44) | -5.1 (13.8)
  Aspartate aminotransferase, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Aspartate aminotransferase, Week 36, n= 219, 204 | -6.4 (31.42) | -6.5 (16.63)
  Aspartate aminotransferase, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Aspartate aminotransferase, Week 48, n= 208, 192 | -7.5 (22.19) | -3.7 (25.28)
  Creatine Kinase, Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Creatine Kinase, Week 4, n= 245, 237 | -0.3 (68.72) | 35.6 (549.1)
  Creatine Kinase, Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Creatine Kinase, Week 12, n= 236, 226 | 6.9 (73.7) | 7.3 (90.39)
  Creatine Kinase, Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Creatine Kinase, Week 24, n= 225, 212 | 10.3 (88.66) | 5.8 (77.12)
  Creatine Kinase, Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Creatine Kinase, Week 36, n= 219, 204 | 11.9 (155.68) | 7.2 (132.74)
  Creatine Kinase, Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Creatine Kinase, Week 48, n= 208, 192 | 23.8 (242.66) | 3.8 (98.58)

16. Secondary Outcome: Change From Baseline in Creatinine Clearance at Indicated Time Points
Description: Clinical chemistry parameters were assessed at Baseline (Day 1), Week 4, 12, 24, 36 and Week 48. Change from Baseline in creatinine clearance is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliter per minute
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Milliliter per minute
  Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Week 4, n= 245, 237 | -16.3 (15.03) | -7.5 (12.91)
  Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Week 12, n= 236, 226 | -17.3 (17.01) | -7 (23.14)
  Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Week 24, n= 225, 212 | -16.2 (20.36) | -9.1 (16.88)
  Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Week 36, n= 219, 204 | -16.8 (22.35) | -7.5 (17.67)
  Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Week 48, n= 208, 192 | -15.9 (19.62) | -7.7 (18.42)

17. Secondary Outcome: Change From Baseline in Lipase at Indicated Timepoints
Description: Clinical chemistry parameters were assessed at Baseline (Day 1), Week 4, 12, 24, 36 and Week 48. Change from Baseline in lipase is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Units per liter
  Week 4, n= 245, 237: number analyzed (Participants) | 245 | 237
  Week 4, n= 245, 237 | -1.2 (15.06) | -1.3 (15.81)
  Week 12, n= 236, 226: number analyzed (Participants) | 236 | 226
  Week 12, n= 236, 226 | -2.2 (22.74) | -2.1 (29)
  Week 24, n= 225, 212: number analyzed (Participants) | 225 | 212
  Week 24, n= 225, 212 | -6 (21.05) | -6 (18.57)
  Week 36, n= 219, 204: number analyzed (Participants) | 219 | 204
  Week 36, n= 219, 204 | -6.3 (25.62) | -6.3 (21.36)
  Week 48, n= 208, 192: number analyzed (Participants) | 208 | 192
  Week 48, n= 208, 192 | -6.5 (29.63) | -7.8 (20.72)

18. Secondary Outcome: Change From Baseline in Total CHLS/HDL CHLS Ratio at Indicated Timepoints
Description: Clinical chemistry parameters were assessed at Baseline (Day 1), Week 4, 12, 24, 36 and Week 48. Change from Baseline in Total CHLS/HDL CHLS ratio is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Ratio
  Week 4, n= 1, 4: number analyzed (Participants) | 1 | 4
  Week 4, n= 1, 4 | 0.1264 (NA) — NA indicates standard deviation could not be calculated for a single participant | 0.2159 (0.60727)
  Week 12, n= 233, 223: number analyzed (Participants) | 233 | 223
  Week 12, n= 233, 223 | -0.2736 (1.0283) | -0.1092 (0.73776)
  Week 24, n= 224, 209: number analyzed (Participants) | 224 | 209
  Week 24, n= 224, 209 | -0.3098 (1.11093) | -0.1922 (0.79848)
  Week 36, n= 212, 198: number analyzed (Participants) | 212 | 198
  Week 36, n= 212, 198 | -0.3286 (1.01181) | -0.1433 (0.79498)
  Week 48, n= 207, 186: number analyzed (Participants) | 207 | 186
  Week 48, n= 207, 186 | -0.2886 (1.01415) | -0.1444 (1.23362)

19. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes at Indicated Time Points
Description: Hematology parameters were assessed at Baseline (Day 1), Week 4, 12, 24, 36 and Week 48. Change from Baseline in basophils, eosinophils, lymphocytes, monocytes is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
10^9 cells per liter
  Basophils, Week 4, n= 241, 234: number analyzed (Participants) | 241 | 234
  Basophils, Week 4, n= 241, 234 | 0.003 (0.0182) | 0.003 (0.0198)
  Basophils, Week 12, n= 228, 216: number analyzed (Participants) | 228 | 216
  Basophils, Week 12, n= 228, 216 | 0.002 (0.0174) | 0.003 (0.0162)
  Basophils, Week 24, n= 221, 208: number analyzed (Participants) | 221 | 208
  Basophils, Week 24, n= 221, 208 | 0.004 (0.0187) | 0.003 (0.0155)
  Basophils, Week 36, n= 214, 203: number analyzed (Participants) | 214 | 203
  Basophils, Week 36, n= 214, 203 | 0.004 (0.0182) | 0.003 (0.0158)
  Basophils, Week 48, n= 206, 189: number analyzed (Participants) | 206 | 189
  Basophils, Week 48, n= 206, 189 | 0.005 (0.0199) | 0.006 (0.0146)
  Eosinophils, Week 4, n= 241, 234: number analyzed (Participants) | 241 | 234
  Eosinophils, Week 4, n= 241, 234 | 0.040 (0.1486) | 0.021 (0.1648)
  Eosinophils, Week 12, n= 228, 216: number analyzed (Participants) | 228 | 216
  Eosinophils, Week 12, n= 228, 216 | 0.037 (0.1982) | -0.001 (0.1610)
  Eosinophils, Week 24, n= 221, 208: number analyzed (Participants) | 221 | 208
  Eosinophils, Week 24, n= 221, 208 | 0.028 (0.1927) | 0.005 (0.1973)
  Eosinophils, Week 36, n= 214, 203: number analyzed (Participants) | 214 | 203
  Eosinophils, Week 36, n= 214, 203 | 0.048 (0.2244) | 0.014 (0.2139)
  Eosinophils, Week 48, n= 206, 189: number analyzed (Participants) | 206 | 189
  Eosinophils, Week 48, n= 206, 189 | 0.030 (0.1744) | 0.007 (0.2274)
  Lymphocytes, Week 4, n= 241, 234: number analyzed (Participants) | 241 | 234
  Lymphocytes, Week 4, n= 241, 234 | 0.208 (0.4914) | 0.119 (0.5493)
  Lymphocytes, Week 12, n= 228, 216: number analyzed (Participants) | 228 | 216
  Lymphocytes, Week 12, n= 228, 216 | 0.257 (0.5500) | 0.156 (0.6690)
  Lymphocytes, Week 24, n= 221, 208: number analyzed (Participants) | 221 | 208
  Lymphocytes, Week 24, n= 221, 208 | 0.317 (0.4889) | 0.192 (0.5910)
  Lymphocytes, Week 36, n= 214, 203: number analyzed (Participants) | 214 | 203
  Lymphocytes, Week 36, n= 214, 203 | 0.362 (0.5199) | 0.178 (0.6441)
  Lymphocytes, Week 48, n= 206, 189: number analyzed (Participants) | 206 | 189
  Lymphocytes, Week 48, n= 206, 189 | 0.359 (0.5235) | 0.261 (0.7098)
  Monocytes, Week 4, n= 241, 234: number analyzed (Participants) | 241 | 234
  Monocytes, Week 4, n= 241, 234 | -0.001 (0.1558) | -0.015 (0.1391)
  Monocytes, Week 12, n= 228, 216: number analyzed (Participants) | 228 | 216
  Monocytes, Week 12, n= 228, 216 | -0.010 (0.1412) | -0.031 (0.1369)
  Monocytes, Week 24, n= 221, 208: number analyzed (Participants) | 221 | 208
  Monocytes, Week 24, n= 221, 208 | 0.008 (0.1498) | -0.015 (0.1581)
  Monocytes, Week 36, n= 214, 203: number analyzed (Participants) | 214 | 203
  Monocytes, Week 36, n= 214, 203 | -0.006 (0.1448) | -0.028 (0.1500)
  Monocytes, Week 48, n= 206, 189: number analyzed (Participants) | 206 | 189
  Monocytes, Week 48, n= 206, 189 | 0.001 (0.1379) | -0.024 (0.1638)

20. Secondary Outcome: Change From Baseline in Erythrocytes at Indicated Time Points
Description: Hematology parameters were assessed at Baseline (Day 1), Week 4, 12, 24, 36 and Week 48. Change from Baseline in erythrocytes is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
10^12 cells per liter
  Week 4, n= 243, 234: number analyzed (Participants) | 243 | 234
  Week 4, n= 243, 234 | -0.04 (0.244) | -0.07 (0.239)
  Week 12, n= 233, 220: number analyzed (Participants) | 233 | 220
  Week 12, n= 233, 220 | -0.07 (0.351) | -0.09 (0.308)
  Week 24, n= 225, 211: number analyzed (Participants) | 225 | 211
  Week 24, n= 225, 211 | -0.08 (0.373) | -0.09 (0.329)
  Week 36, n= 218, 203: number analyzed (Participants) | 218 | 203
  Week 36, n= 218, 203 | -0.10 (0.384) | -0.08 (0.358)
  Week 48, n= 207, 190: number analyzed (Participants) | 207 | 190
  Week 48, n= 207, 190 | -0.10 (0.365) | -0.05 (0.318)

21. Secondary Outcome: Change From Baseline in Hematocrit Count at Indicated Time Points
Description: Hematology parameters were assessed at Baseline (Day 1), Weeks 4, 12, 24, 36 and 48. Change from Baseline in hematocrit is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Proportion of red blood cells in blood
  Week 4, n= 243, 234: number analyzed (Participants) | 243 | 234
  Week 4, n= 243, 234 | 0.0003 (0.02176) | -0.0042 (0.02238)
  Week 12, n= 233, 220: number analyzed (Participants) | 233 | 220
  Week 12, n= 233, 220 | 0.0081 (0.03157) | 0.0000 (0.02646)
  Week 24, n= 225, 211: number analyzed (Participants) | 225 | 211
  Week 24, n= 225, 211 | 0.0157 (0.03209) | 0.0051 (0.03083)
  Week 36, n= 218, 203: number analyzed (Participants) | 218 | 203
  Week 36, n= 218, 203 | 0.0167 (0.03451) | 0.0062 (0.03379)
  Week 48, n= 207, 190: number analyzed (Participants) | 207 | 190
  Week 48, n= 207, 190 | 0.0212 (0.03293) | 0.0107 (0.03200)

22. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume at Indicated Time Points
Description: Hematology parameters were assessed at Baseline (Day 1), Week 4, 12, 24, 36 and Week 48. Change from Baseline in erythrocyte mean corpuscular volume (EMCV) is summarized. Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 4, Week 12, Week 24, Week 36 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Femtoliter
  Week 4, n= 243, 234: number analyzed (Participants) | 243 | 234
  Week 4, n= 243, 234 | 0.9 (1.81) | 0.5 (1.83)
  Week 12, n= 233, 220: number analyzed (Participants) | 233 | 220
  Week 12, n= 233, 220 | 3.4 (2.98) | 1.9 (2.94)
  Week 24, n= 225, 211: number analyzed (Participants) | 225 | 211
  Week 24, n= 225, 211 | 5.5 (4.03) | 3.1 (4.33)
  Week 36, n= 218, 203: number analyzed (Participants) | 218 | 203
  Week 36, n= 218, 203 | 6.0 (4.04) | 3.1 (5.22)
  Week 48, n= 207, 190: number analyzed (Participants) | 207 | 190
  Week 48, n= 207, 190 | 7.1 (4.31) | 3.7 (5.15)

23. Secondary Outcome: Change From Baseline in Triglycerides at Week 48
Description: Change from Baseline in mean triglycerides is summarized at Week 48. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value. Adjusted mean is the estimated mean change from Baseline in fasted triglycerides at Week 48 in each arm calculated from a model adjusted for the following covariates: treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age and triglycerides at Baseline. Participants on lipid lowering therapy at Baseline were excluded from analysis. Measurements collected after a participant initiates lipid lowering therapy were set to missing. Missing values were imputed using multiple imputation under a multivariate normal model adjusting for Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, fasted triglycerides and TC/HDL ratio at Baseline, Week 12 and Week 36.
Time Frame: Baseline (Day 1) and Week 48
Population: Safety Population. Participants on lipid lowering therapy at Baseline were excluded from analysis. Only those participants with data available at specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 226 | 214
Millimoles per liter | 0.045 (0.0477) | 0.070 (0.0477)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p = 0.7053, Multiple Imputed Dataset - MAR; Mean Difference (Final Values) = -0.026, 95% CI 2-sided [-0.159 to 0.107]

24. Secondary Outcome: Change From Baseline in TC/HDL Ratio at Week 48
Description: Change from Baseline in mean total cholesterol (TC)/HDL ratio is summarized at Week 48. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value. Adjusted mean is the estimated mean change from Baseline in fasted TC/HDL at Week 48 in each arm calculated from a model adjusted for the following covariates: treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age and triglycerides/HDL at Baseline. Participants on lipid lowering therapy at Baseline were excluded from analysis. Measurements collected after a participant initiates lipid lowering therapy were set to missing. Missing values were imputed using multiple imputation under a multivariate normal model adjusting for Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, fasted triglycerides and TC/HDL ratio at Baseline, Week 12 and Week 36.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 226 | 214
Ratio | -0.264 (0.0707) | -0.158 (0.0784)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p = 0.3165, Multiple Imputed Dataset - MAR; Mean Difference (Final Values) = -0.106, 95% CI 2-sided [-0.313 to 0.101]

25. Secondary Outcome: Change From Baseline in Urine Albumin Creatinine Ratio at Indicated Time Points
Description: Change from Baseline in urine albumin creatinine ratio at Week 24 and Week 48 is summarized. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milligrams per millimole
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
milligrams per millimole
  Week 24, n= 179, 186: number analyzed (Participants) | 179 | 186
  Week 24, n= 179, 186 | -1.15 (16.557) | -1.03 (9.091)
  Week 48, n= 170, 164: number analyzed (Participants) | 170 | 164
  Week 48, n= 170, 164 | -0.68 (20.597) | -0.10 (9.393)

26. Secondary Outcome: Number of Participants With AEs by Maximum Toxicity-Randomized Phase
Description: Number of participants with Grade 1-4 AEs by maximum toxicity were assessed from the start of study treatment and until end of the Randomization phase. AEs are categorized into following grades as per The Division of Aqcuired Immuno Deficiency Syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table)- Grade 1- mild, Grade 2- moderate; Grade 3- severe and Grade 4- potentially life-threatening. Higher the grade, more severe the symptoms.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Participants
  Grade 1 | 79 | 60
  Grade 2 | 94 | 91
  Grade 3 | 18 | 37
  Grade 4 | 3 | 9

27. Secondary Outcome: Number of Participants With AEs by Maximum Toxicity-Continuation Phase
Description: Number of participants with Grade 1-4 AEs were assessed in Continuation Phase. AEs are categorized into following grades as per The Division of Aqcuired Immuno Deficiency Syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table)- Grade 1- mild, Grade 2- moderate; Grade 3- severe and Grade 4- potentially life-threatening. Higher the grade, more severe the symptoms.
Time Frame: From Weeks 48 to 432
Population: Safety - Continuation Phase Population comprised of all participants in the DTG/ABC/3TC group who received at least 1 dose of study treatment after entering the Continuation Phase
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Participants
  Grade 1 | 32
  Grade 2 | 48
  Grade 3 | 7
  Grade 4 | 6

28. Secondary Outcome: Number of Participants With Any Adverse Events (AEs), and Serious Adverse Events (SAEs)-Randomized Phase
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or other events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcome listed above, liver injury and impaired liver function and grade 4 laboratory abnormalities. Number of participants with any AEs, and SAEs have been presented.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Participants
  Any AEs | 195 | 197
  Any SAEs | 12 | 20

29. Secondary Outcome: Number of Participants With Any AEs, and SAEs in Continuation Phase
Description: as for outcome 28
Time Frame: From Weeks 48 to 432
Population: Safety-Continuation Phase Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Participants
  Any AEs | 93
  Any SAEs | 13

30. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Chemistry Toxicities-Randomized Phase
Description: Number of participants with Grade 1-4 emergent chemistry toxicities were assessed from the start of study treatment and end of Randomized Phase. Chemistry toxicities were categorized into following grades as per The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table)- Grade 1- mild, Grade 2- moderate; Grade 3- severe and Grade 4- potentially life-threatening. Higher the grade, more severe the symptoms. Data has been reported for clinical chemistry parameters including hyperglycaemia, hyperkalemia, hypernatremia, hypoglycaemia, hypokalemia, hyponatremia, alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, carbon dioxide, cholesterol, creatine kinase, creatinine, LDL cholesterol calculation, LDL cholesterol direct, lipase, phosphate, potassium, sodium, triglycerides and glucose.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Participants
  Hyperglycaemia, Grade 1 | 17 | 11
  Hyperglycaemia, Grade 2 | 16 | 9
  Hyperglycaemia, Grade 3 | 4 | 3
  Hyperglycaemia, Grade 4 | 1 | 0
  Hyperkalemia, Grade 1 | 1 | 0
  Hyperkalemia, Grade 2 | 0 | 1
  Hyperkalemia, Grade 3 | 0 | 0
  Hyperkalemia, Grade 4 | 0 | 0
  Hypernatremia, Grade 1 | 1 | 0
  Hypernatremia, Grade 2 | 0 | 0
  Hypernatremia, Grade 3 | 0 | 0
  Hypernatremia, Grade 4 | 0 | 0
  Hypoglycaemia, Grade 1 | 6 | 5
  Hypoglycaemia, Grade 2 | 3 | 1
  Hypoglycaemia, Grade 3 | 1 | 0
  Hypoglycaemia, Grade 4 | 0 | 0
  Hypokalemia, Grade 1 | 17 | 19
  Hypokalemia, Grade 2 | 1 | 0
  Hypokalemia, Grade 3 | 0 | 0
  Hypokalemia, Grade 4 | 0 | 0
  Hyponatremia, Grade 1 | 44 | 57
  Hyponatremia, Grade 2 | 1 | 0
  Hyponatremia, Grade 3 | 0 | 0
  Hyponatremia, Grade 4 | 0 | 0
  Alanine aminotransferase, Grade 1 | 5 | 7
  Alanine aminotransferase, Grade 2 | 6 | 4
  Alanine aminotransferase, Grade 3 | 1 | 2
  Alanine aminotransferase, Grade 4 | 1 | 0
  Albumin, Grade 1 | 3 | 2
  Albumin, Grade 2 | 0 | 2
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  Alkaline phosphatase, Grade 1 | 3 | 14
  Alkaline phosphatase, Grade 2 | 2 | 1
  Alkaline phosphatase, Grade 3 | 0 | 0
  Alkaline phosphatase, Grade 4 | 0 | 0
  Aspartate aminotransferase, Grade 1 | 12 | 7
  Aspartate aminotransferase, Grade 2 | 4 | 4
  Aspartate aminotransferase, Grade 3 | 1 | 2
  Aspartate aminotransferase, Grade 4 | 1 | 0
  Bilirubin, Grade 1 | 2 | 52
  Bilirubin, Grade 2 | 0 | 86
  Bilirubin, Grade 3 | 0 | 57
  Bilirubin, Grade 4 | 0 | 5
  Carbon dioxide, Grade 1 | 65 | 54
  Carbon dioxide, Grade 2 | 4 | 3
  Carbon dioxide, Grade 3 | 0 | 0
  Carbon dioxide, Grade 4 | 0 | 0
  Cholesterol, Grade 1 | 52 | 31
  Cholesterol, Grade 2 | 28 | 9
  Cholesterol, Grade 3 | 4 | 2
  Cholesterol, Grade 4 | 0 | 0
  Creatine kinase, Grade 1 | 3 | 5
  Creatine kinase, Grade 2 | 1 | 1
  Creatine kinase, Grade 3 | 3 | 0
  Creatine kinase, Grade 4 | 0 | 1
  Creatinine, Grade 1 | 3 | 7
  Creatinine, Grade 2 | 0 | 3
  Creatinine, Grade 3 | 1 | 0
  Creatinine, Grade 4 | 0 | 0
  LDL cholesterol calculation, Grade 1 | 38 | 21
  LDL cholesterol calculation, Grade 2 | 13 | 9
  LDL cholesterol calculation, Grade 3 | 7 | 2
  LDL cholesterol calculation, Grade 4 | 0 | 0
  LDL cholesterol direct, Grade 1 | 3 | 1
  LDL cholesterol direct, Grade 2 | 1 | 0
  LDL cholesterol direct, Grade 3 | 0 | 0
  LDL cholesterol direct, Grade 4 | 0 | 0
  Lipase, Grade 1 | 12 | 7
  Lipase, Grade 2 | 5 | 3
  Lipase, Grade 3 | 3 | 2
  Lipase, Grade 4 | 0 | 1
  Phosphate, Grade 1 | 5 | 11
  Phosphate, Grade 2 | 7 | 9
  Phosphate, Grade 3 | 1 | 2
  Phosphate, Grade 4 | 0 | 0
  Potassium, Grade 1 | 18 | 19
  Potassium, Grade 2 | 1 | 1
  Potassium, Grade 3 | 0 | 0
  Potassium, Grade 4 | 0 | 0
  Sodium, Grade 1 | 45 | 57
  Sodium, Grade 2 | 1 | 0
  Sodium, Grade 3 | 0 | 0
  Sodium, Grade 4 | 0 | 0
  Triglycerides, Grade 1 | 0 | 0
  Triglycerides, Grade 2 | 5 | 2
  Triglycerides, Grade 3 | 2 | 0
  Triglycerides, Grade 4 | 0 | 0
  Glucose, Grade 1 | 22 | 15
  Glucose, Grade 2 | 19 | 10
  Glucose, Grade 3 | 4 | 3
  Glucose, Grade 4 | 1 | 0

31. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Chemistry Toxicities-Continuation Phase
Description: Number of participants with grades 1-4 emergent chemistry toxicities were assessed in Continuation Phase. Chemistry toxicities were categorized into following grades as per The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table)- Grade 1- mild, Grade 2- moderate; Grade 3- severe and Grade 4- potentially life-threatening. Higher the grade, more severe the symptoms. Data has been reported for clinical chemistry parameters including hyperglycaemia, hypernatremia, hypoglycaemia, hypokalemia, hyponatremia, alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bilirubin, carbon dioxide, cholesterol, creatine kinase, creatinine, LDL cholesterol calculation, LDL cholesterol direct, lipase, phosphate, potassium, sodium, triglycerides and glucose.
Time Frame: From Weeks 48 to 432
Population: Safety - Continuation Phase Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Participants
  Hyperglycaemia, Grade 1, n=143: number analyzed (Participants) | 143
  Hyperglycaemia, Grade 1, n=143 | 24
  Hyperglycaemia, Grade 2, n=143: number analyzed (Participants) | 143
  Hyperglycaemia, Grade 2, n=143 | 9
  Hyperglycaemia, Grade 3, n=143: number analyzed (Participants) | 143
  Hyperglycaemia, Grade 3, n=143 | 3
  Hyperglycaemia, Grade 4, n=143: number analyzed (Participants) | 143
  Hyperglycaemia, Grade 4, n=143 | 0
  Hypernatremia, Grade 1, n=146: number analyzed (Participants) | 146
  Hypernatremia, Grade 1, n=146 | 2
  Hypernatremia, Grade 2, n=146: number analyzed (Participants) | 146
  Hypernatremia, Grade 2, n=146 | 0
  Hypernatremia, Grade 3, n=146: number analyzed (Participants) | 146
  Hypernatremia, Grade 3, n=146 | 0
  Hypernatremia, Grade 4, n=146: number analyzed (Participants) | 146
  Hypernatremia, Grade 4, n=146 | 0
  Hypoglycaemia, Grade 1, n=143: number analyzed (Participants) | 143
  Hypoglycaemia, Grade 1, n=143 | 1
  Hypoglycaemia, Grade 2, n=143: number analyzed (Participants) | 143
  Hypoglycaemia, Grade 2, n=143 | 0
  Hypoglycaemia, Grade 3, n=143: number analyzed (Participants) | 143
  Hypoglycaemia, Grade 3, n=143 | 0
  Hypoglycaemia, Grade 4, n=143: number analyzed (Participants) | 143
  Hypoglycaemia, Grade 4, n=143 | 1
  Hypokalemia, Grade 1, n=146: number analyzed (Participants) | 146
  Hypokalemia, Grade 1, n=146 | 13
  Hypokalemia, Grade 2, n=146: number analyzed (Participants) | 146
  Hypokalemia, Grade 2, n=146 | 0
  Hypokalemia, Grade 3, n=146: number analyzed (Participants) | 146
  Hypokalemia, Grade 3, n=146 | 0
  Hypokalemia, Grade 4, n=146: number analyzed (Participants) | 146
  Hypokalemia, Grade 4, n=146 | 0
  Hyponatremia, Grade 1, n=146: number analyzed (Participants) | 146
  Hyponatremia, Grade 1, n=146 | 36
  Hyponatremia, Grade 2, n=146: number analyzed (Participants) | 146
  Hyponatremia, Grade 2, n=146 | 0
  Hyponatremia, Grade 3, n=146: number analyzed (Participants) | 146
  Hyponatremia, Grade 3, n=146 | 0
  Hyponatremia, Grade 4, n=146: number analyzed (Participants) | 146
  Hyponatremia, Grade 4, n=146 | 0
  Alanine aminotransferase, Grade 1, n=146: number analyzed (Participants) | 146
  Alanine aminotransferase, Grade 1, n=146 | 7
  Alanine aminotransferase, Grade 2, n=146: number analyzed (Participants) | 146
  Alanine aminotransferase, Grade 2, n=146 | 3
  Alanine aminotransferase, Grade 3, n=146: number analyzed (Participants) | 146
  Alanine aminotransferase, Grade 3, n=146 | 0
  Alanine aminotransferase, Grade 4, n=146: number analyzed (Participants) | 146
  Alanine aminotransferase, Grade 4, n=146 | 2
  Alkaline phosphatase, Grade 1, n=146: number analyzed (Participants) | 146
  Alkaline phosphatase, Grade 1, n=146 | 5
  Alkaline phosphatase, Grade 2, n=146: number analyzed (Participants) | 146
  Alkaline phosphatase, Grade 2, n=146 | 0
  Alkaline phosphatase, Grade 3, n=146: number analyzed (Participants) | 146
  Alkaline phosphatase, Grade 3, n=146 | 0
  Alkaline phosphatase, Grade 4, n=146: number analyzed (Participants) | 146
  Alkaline phosphatase, Grade 4, n=146 | 0
  Aspartate aminotransferase, Grade 1, n=146: number analyzed (Participants) | 146
  Aspartate aminotransferase, Grade 1, n=146 | 10
  Aspartate aminotransferase, Grade 2, n=146: number analyzed (Participants) | 146
  Aspartate aminotransferase, Grade 2, n=146 | 2
  Aspartate aminotransferase, Grade 3, n=146: number analyzed (Participants) | 146
  Aspartate aminotransferase, Grade 3, n=146 | 0
  Aspartate aminotransferase, Grade 4, n=146: number analyzed (Participants) | 146
  Aspartate aminotransferase, Grade 4, n=146 | 2
  Bilirubin, Grade 1, n=146: number analyzed (Participants) | 146
  Bilirubin, Grade 1, n=146 | 4
  Bilirubin, Grade 2, n=146: number analyzed (Participants) | 146
  Bilirubin, Grade 2, n=146 | 1
  Bilirubin, Grade 3, n=146: number analyzed (Participants) | 146
  Bilirubin, Grade 3, n=146 | 3
  Bilirubin, Grade 4, n=146: number analyzed (Participants) | 146
  Bilirubin, Grade 4, n=146 | 0
  Carbon dioxide, Grade 1, n=146: number analyzed (Participants) | 146
  Carbon dioxide, Grade 1, n=146 | 58
  Carbon dioxide, Grade 2, n=146: number analyzed (Participants) | 146
  Carbon dioxide, Grade 2, n=146 | 7
  Carbon dioxide, Grade 3, n=146: number analyzed (Participants) | 146
  Carbon dioxide, Grade 3, n=146 | 0
  Carbon dioxide, Grade 4, n=146: number analyzed (Participants) | 146
  Carbon dioxide, Grade 4, n=146 | 0
  Cholesterol, Grade 1, n=71: number analyzed (Participants) | 71
  Cholesterol, Grade 1, n=71 | 9
  Cholesterol, Grade 2, n=71: number analyzed (Participants) | 71
  Cholesterol, Grade 2, n=71 | 9
  Cholesterol, Grade 3, n=71: number analyzed (Participants) | 71
  Cholesterol, Grade 3, n=71 | 3
  Cholesterol, Grade 4, n=71: number analyzed (Participants) | 71
  Cholesterol, Grade 4, n=71 | 0
  Creatine kinase, Grade 1, n=146: number analyzed (Participants) | 146
  Creatine kinase, Grade 1, n=146 | 6
  Creatine kinase, Grade 2, n=146: number analyzed (Participants) | 146
  Creatine kinase, Grade 2, n=146 | 1
  Creatine kinase, Grade 3, n=146: number analyzed (Participants) | 146
  Creatine kinase, Grade 3, n=146 | 1
  Creatine kinase, Grade 4, n=146: number analyzed (Participants) | 146
  Creatine kinase, Grade 4, n=146 | 1
  Creatinine, Grade 1, n=146: number analyzed (Participants) | 146
  Creatinine, Grade 1, n=146 | 5
  Creatinine, Grade 2, n=146: number analyzed (Participants) | 146
  Creatinine, Grade 2, n=146 | 0
  Creatinine, Grade 3, n=146: number analyzed (Participants) | 146
  Creatinine, Grade 3, n=146 | 0
  Creatinine, Grade 4, n=146: number analyzed (Participants) | 146
  Creatinine, Grade 4, n=146 | 1
  LDL cholesterol calculation, Grade 1, n=70: number analyzed (Participants) | 70
  LDL cholesterol calculation, Grade 1, n=70 | 5
  LDL cholesterol calculation, Grade 2, n=70: number analyzed (Participants) | 70
  LDL cholesterol calculation, Grade 2, n=70 | 8
  LDL cholesterol calculation, Grade 3, n=70: number analyzed (Participants) | 70
  LDL cholesterol calculation, Grade 3, n=70 | 2
  LDL cholesterol calculation, Grade 4, n=70: number analyzed (Participants) | 70
  LDL cholesterol calculation, Grade 4, n=70 | 0
  LDL cholesterol direct, Grade 1, n=2: number analyzed (Participants) | 2
  LDL cholesterol direct, Grade 1, n=2 | 1
  LDL cholesterol direct, Grade 2, n=2: number analyzed (Participants) | 2
  LDL cholesterol direct, Grade 2, n=2 | 0
  LDL cholesterol direct, Grade 3, n=2: number analyzed (Participants) | 2
  LDL cholesterol direct, Grade 3, n=2 | 0
  LDL cholesterol direct, Grade 4, n=2: number analyzed (Participants) | 2
  LDL cholesterol direct, Grade 4, n=2 | 0
  Lipase, Grade 1, n=146: number analyzed (Participants) | 146
  Lipase, Grade 1, n=146 | 9
  Lipase, Grade 2, n=146: number analyzed (Participants) | 146
  Lipase, Grade 2, n=146 | 6
  Lipase, Grade 3, n=146: number analyzed (Participants) | 146
  Lipase, Grade 3, n=146 | 1
  Lipase, Grade 4, n=146: number analyzed (Participants) | 146
  Lipase, Grade 4, n=146 | 1
  Phosphate, Grade 1, n=146: number analyzed (Participants) | 146
  Phosphate, Grade 1, n=146 | 2
  Phosphate, Grade 2, n=146: number analyzed (Participants) | 146
  Phosphate, Grade 2, n=146 | 15
  Phosphate, Grade 3, n=146: number analyzed (Participants) | 146
  Phosphate, Grade 3, n=146 | 2
  Phosphate, Grade 4, n=146: number analyzed (Participants) | 146
  Phosphate, Grade 4, n=146 | 0
  Potassium, Grade 1, n=146: number analyzed (Participants) | 146
  Potassium, Grade 1, n=146 | 13
  Potassium, Grade 2, n=146: number analyzed (Participants) | 146
  Potassium, Grade 2, n=146 | 0
  Potassium, Grade 3, n=146: number analyzed (Participants) | 146
  Potassium, Grade 3, n=146 | 0
  Potassium, Grade 4, n=146: number analyzed (Participants) | 146
  Potassium, Grade 4, n=146 | 0
  Sodium, Grade 1, n=146: number analyzed (Participants) | 146
  Sodium, Grade 1, n=146 | 37
  Sodium, Grade 2, n=146: number analyzed (Participants) | 146
  Sodium, Grade 2, n=146 | 0
  Sodium, Grade 3, n=146: number analyzed (Participants) | 146
  Sodium, Grade 3, n=146 | 0
  Sodium, Grade 4, n=146: number analyzed (Participants) | 146
  Sodium, Grade 4, n=146 | 0
  Triglycerides, Grade 1, n=71: number analyzed (Participants) | 71
  Triglycerides, Grade 1, n=71 | 0
  Triglycerides, Grade 2, n=71: number analyzed (Participants) | 71
  Triglycerides, Grade 2, n=71 | 1
  Triglycerides, Grade 3, n=71: number analyzed (Participants) | 71
  Triglycerides, Grade 3, n=71 | 0
  Triglycerides, Grade 4, n=71: number analyzed (Participants) | 71
  Triglycerides, Grade 4, n=71 | 0
  Glucose, Grade 1, n=143: number analyzed (Participants) | 143
  Glucose, Grade 1, n=143 | 24
  Glucose, Grade 2, n=143: number analyzed (Participants) | 143
  Glucose, Grade 2, n=143 | 9
  Glucose, Grade 3, n=143: number analyzed (Participants) | 143
  Glucose, Grade 3, n=143 | 3
  Glucose, Grade 4, n=143: number analyzed (Participants) | 143
  Glucose, Grade 4, n=143 | 1

32. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities-Randomized Phase
Description: Number of participants with Grade 1-4 emergent hematology toxicities were assessed from the start of study treatment and end of Randomized Phase. Hematology toxicities were categorized into following grades as per The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table)- Grade 1- mild, Grade 2- moderate; Grade 3- severe and Grade 4- potentially life-threatening. Higher the grade, more severe the symptoms. Data has been reported for clinical chemistry parameters including hemoglobin, leukocytes, neutrophils and platelets.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Participants
  Hemoglobin, Grade 1 | 7 | 21
  Hemoglobin, Grade 2 | 2 | 3
  Hemoglobin, Grade 3 | 1 | 1
  Hemoglobin, Grade 4 | 0 | 0
  Leukocytes, Grade 1 | 5 | 6
  Leukocytes, Grade 2 | 1 | 2
  Leukocytes, Grade 3 | 0 | 0
  Leukocytes, Grade 4 | 0 | 0
  Neutrophils, Grade 1 | 15 | 12
  Neutrophils, Grade 2 | 7 | 9
  Neutrophils, Grade 3 | 0 | 2
  Neutrophils, Grade 4 | 1 | 1
  Platelets, Grade 1 | 6 | 1
  Platelets, Grade 2 | 0 | 2
  Platelets, Grade 3 | 1 | 0
  Platelets, Grade 4 | 0 | 0

33. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities-Continuation Phase
Description: Number of participants with Grade 1-4 emergent hematology toxicities were assessed in Continuation Phase. Hematology toxicities were categorized into following grades as per The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table)- Grade 1- mild, Grade 2- moderate; Grade 3- severe and Grade 4- potentially life-threatening. Higher the grade, more severe the symptoms. Data has been reported for clinical chemistry parameters including hemoglobin, leukocytes, neutrophils and platelets.
Time Frame: From Weeks 48 to 432
Population: Safety - Continuation Phase Population. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 146
Participants
  Hemoglobin, Grade 1 | 5
  Hemoglobin, Grade 2 | 1
  Hemoglobin, Grade 3 | 0
  Hemoglobin, Grade 4 | 0
  Leukocytes, Grade 1 | 2
  Leukocytes, Grade 2 | 0
  Leukocytes, Grade 3 | 1
  Leukocytes, Grade 4 | 0
  Neutrophils, Grade 1 | 10
  Neutrophils, Grade 2 | 2
  Neutrophils, Grade 3 | 1
  Neutrophils, Grade 4 | 1
  Platelets, Grade 1 | 3
  Platelets, Grade 2 | 1
  Platelets, Grade 3 | 0
  Platelets, Grade 4 | 0

34. Secondary Outcome: Number of Participants Who Withdrew From Treatment Due to AEs-Randomized Phase
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of an MP. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is an important medical event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or is associated with liver injury and impaired liver function.
Time Frame: Up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Participants | 10 | 17

35. Secondary Outcome: Number of Participants Who Withdrew From Treatment Due to AEs-Continuation Phase
Description: as for outcome 34
Time Frame: From Weeks 48 to 432
Population: Safety - Continuation Phase Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
Number analyzed (Participants) | 149
Participants | 4

36. Secondary Outcome: Change From Baseline in Bone Specific Alkaline Phosphatase, Osteocalcin and Procollagen 1 N-terminal Propeptide at Indicated Timepoints
Description: Bone markers were assessed at Baseline (Day 1), Weeks 24, 48. Change from Baseline in bone specific alkaline phosphatase (BSAP), osteocalcin and procollagen 1 N-terminal propeptide (PTP) is summarized. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Micrograms per liter
  BSAP, Week 24, n=219, 207: number analyzed (Participants) | 219 | 207
  BSAP, Week 24, n=219, 207 | 1.33 (3.934) | 6.00 (5.962)
  BSAP, Week 48, n=202, 184: number analyzed (Participants) | 202 | 184
  BSAP, Week 48, n=202, 184 | 2.64 (5.746) | 7.60 (7.144)
  Osteocalcin, Week 24, n=209, 197: number analyzed (Participants) | 209 | 197
  Osteocalcin, Week 24, n=209, 197 | 3.73 (7.484) | 14.38 (22.205)
  Osteocalcin, Week 48, n=194, 178: number analyzed (Participants) | 194 | 178
  Osteocalcin, Week 48, n=194, 178 | 5.15 (9.018) | 16.30 (25.043)
  PTP, Week 24, n=223, 206: number analyzed (Participants) | 223 | 206
  PTP, Week 24, n=223, 206 | 10.1 (20.11) | 32.0 (27.89)
  PTP, Week 48, n=205, 186: number analyzed (Participants) | 205 | 186
  PTP, Week 48, n=205, 186 | 11.2 (23.05) | 34.1 (27.28)

37. Secondary Outcome: Change From Baseline in Type I Collagen C-telopeptides at Indicated Timepoints
Description: Bone markers were assessed at Baseline (Day 1), Weeks 24, 48. Change from Baseline in Type I collagen C-telopeptides (T-1 CCT) is summarized. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Nanograms per liter
  Week 24, n=221, 207: number analyzed (Participants) | 221 | 207
  Week 24, n=221, 207 | 89.8 (173.09) | 272.4 (205.22)
  Week 48, n=202, 185: number analyzed (Participants) | 202 | 185
  Week 48, n=202, 185 | 75.9 (173.73) | 267.9 (200.82)

38. Secondary Outcome: Change From Baseline in Vitamin D, Vitamin D2 and Vitamin D3 at Week 24 and Week 48
Description: Bone markers were assessed at Baseline (Day 1), Weeks 24, 48. Change from Baseline in vitamin D, vitamin D2 and vitamin D3 is summarized. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Weeks 24 and 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Nanomoles per liter
  Vitamin D, Week 24, n=223, 208: number analyzed (Participants) | 223 | 208
  Vitamin D, Week 24, n=223, 208 | 1.8 (24.95) | 16.3 (31.66)
  Vitamin D, Week 48, n=206, 186: number analyzed (Participants) | 206 | 186
  Vitamin D, Week 48, n=206, 186 | -1.9 (20.63) | 8.9 (23.78)
  Vitamin D2, Week 24, n=223, 208: number analyzed (Participants) | 223 | 208
  Vitamin D2, Week 24, n=223, 208 | 0.3 (6.04) | 1.0 (7.88)
  Vitamin D2, Week 48, n=206, 186: number analyzed (Participants) | 206 | 186
  Vitamin D2, Week 48, n=206, 186 | 0.1 (4.71) | 0.9 (11.00)
  Vitamin D3, Week 24, n=223, 208: number analyzed (Participants) | 223 | 208
  Vitamin D3, Week 24, n=223, 208 | 1.5 (24.33) | 15.2 (31.39)
  Vitamin D3, Week 48, n=206, 186: number analyzed (Participants) | 206 | 186
  Vitamin D3, Week 48, n=206, 186 | -1.9 (20.56) | 7.9 (21.72)

39. Secondary Outcome: Bone Specific Alkaline Phosphatase, Osteocalcin, Procollagen 1 N-terminal Propeptide, Type 1 Collagen C-Telopeptide, Vitamin D Ratio of Week 48 Results Over Baseline
Description: Bone markers were assessed at indicated timepoints. Bone specific alkaline phosphatase (BSAP), osteocalcin and procollagen 1 N-terminal propeptide (PTP), Type 1 Collagen C-Telopeptide, vitamin D ratio of Week 48 results over Baseline is calculated. Bone biomarkers were analyzed based on log transformed data. Estimates of adjusted mean and difference were calculated from an Analysis of covariance (ANCOVA) model adjusting for age, baseline viral load Baseline CD4+ cell count, Baseline biomarker level, body mass index category, smoking status and baseline Vitamin D use. Adjusted mean of log-transformed change from Baseline are transformed back to Week 48/Baseline ratio for each treatment group. Adjusted difference of log-transformed change from Baseline between treatment groups is transformed back to the ratio of Week 48/Baseline ratio in DTG/ABC/3TC FDC to ATV+RTV+TDF/FTC FDC.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Ratio
  BSAP, n=202, 183: number analyzed (Participants) | 202 | 183
  BSAP, n=202, 183 | 1.188 [1.135 to 1.243] | 1.629 [1.553 to 1.708]
  PTP, n=202, 184: number analyzed (Participants) | 202 | 184
  PTP, n=202, 184 | 1.214 [1.158 to 1.272] | 1.752 [1.668 to 1.840]
  Osteocalcin, n=194, 178: number analyzed (Participants) | 194 | 178
  Osteocalcin, n=194, 178 | 1.282 [1.214 to 1.354] | 2.039 [1.926 to 2.159]
  Type 1 Collagen C-Telopeptide, n=202, 184: number analyzed (Participants) | 202 | 184
  Type 1 Collagen C-Telopeptide, n=202, 184 | 1.257 [1.195 to 1.323] | 1.918 [1.819 to 2.023]
  Vitamin D, n=206, 186: number analyzed (Participants) | 206 | 186
  Vitamin D, n=206, 186 | 0.987 [0.940 to 1.036] | 1.158 [1.101 to 1.219]
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of ratio = 0.729, 95% CI 2-sided [0.683 to 0.779] — BSAP ratio of Week 48 result over Baseline
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of ratio = 0.693, 95% CI 2-sided [0.647 to 0.741] — PTP ratio of Week 48 result over Baseline
Statistical Analysis 3: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p < 0.001, ANCOVA; Ratio of ratio = 0.629, 95% CI 2-sided [0.581 to 0.680] — Osteocalcin ratio of Week 48 result over Baseline
Statistical Analysis 4: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p < 0.0001, ANCOVA; Ratio of ratio = 0.655, 95% CI 2-sided [0.609 to 0.706] — Type 1 Collagen C-Telopeptide ratio of Week 48 result over Baseline
Statistical Analysis 5: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p < 0.0001, ANCOVA; Ratio of ratio = 0.852, 95% CI 2-sided [0.794 to 0.914] — Vitamin D ratio of Week 48 result over Baseline

40. Secondary Outcome: Change From Baseline at Week 48 in SF-12 Total Score, MCS and PCS
Description: The 12-Item Short Form Health Survey (SF-12) is 12 item abbreviated form of SF-36 survey. SF-12 questions make up 8 scales: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, Mental Health. SF-12 is a self-reported outcome measure assessing psychological wellness and the impact of health on an individual's everyday life. SF-12 total score ranges from 20 to 60 and higher score indicate a higher level of functioning. SF-12 total score was calculated by a clinician scoring 12-question survey filled by participants. Transformed physical component summary score (PCS) and transformed mental component summary score (MCS) are derived using the sum of all 12 items and scored onto a 0-100 scale such that a higher score indicates a better health state and better functioning. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Score on a scale
  Total Score, Week 48, n=205, 192: number analyzed (Participants) | 205 | 192
  Total Score, Week 48, n=205, 192 | 0.0 (5.15) | 0.1 (5.66)
  MCS, Week 48, n=205, 192: number analyzed (Participants) | 205 | 192
  MCS, Week 48, n=205, 192 | 2.397 (10.5232) | 2.329 (9.9782)
  PCS, Week 48, n=205, 192: number analyzed (Participants) | 205 | 192
  PCS, Week 48, n=205, 192 | 1.905 (8.6309) | 1.444 (8.3938)

41. Secondary Outcome: HIVTSQs Total Score at Indicated Timepoints
Description: The HIV treatment satisfaction questionnaire (HIVTSQ) is a 10-item self-reported scale that measures overall satisfaction with treatment and by specific domains e.g. convenience, flexibility. The HIVTSQ items are summed up to produce a treatment satisfaction total score (0 to 60) and an individual satisfaction rating for each item (0 to 6) and two subscales: general satisfaction/clinical and lifestyle/ease subscales. The higher the score, the greater the improvement in treatment satisfaction as compared to the past few weeks. A smaller score represents a decline in treatment satisfaction compared to the past few weeks. Statistical analysis was performed based on Wilcoxon rank sum test.
Time Frame: Weeks 4, 12, 24 and 48
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Score on a scale
  Week 4, n=243, 239: number analyzed (Participants) | 243 | 239
  Week 4, n=243, 239 | 54.0 (6.37) | 51.9 (8.53)
  Week 12, n=236, 226: number analyzed (Participants) | 236 | 226
  Week 12, n=236, 226 | 56.1 (5.38) | 53.6 (7.67)
  Week 24, n=225, 211: number analyzed (Participants) | 225 | 211
  Week 24, n=225, 211 | 56.8 (4.55) | 54.3 (7.27)
  Week 48, n=206, 191: number analyzed (Participants) | 206 | 191
  Week 48, n=206, 191 | 57.0 (4.38) | 55.4 (6.00)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney) — Week 4
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Week 12
Statistical Analysis 3: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — Week 24
Statistical Analysis 4: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase vs ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney) — Week 48

42. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/mL at Week 48 by Subgroups
Description: Percentage of participants with plasma HIV-1 RNA <50 copies/mL at Week 48 by subgroups (age, race, country, Baseline plasma HIV-1 RNA [BPHR], Baseline CD4+ cell count [BCCC], Baseline Centers for Disease Control and Prevention [CDC] category and HIV-1 subtype) were assessed using the Snapshot algorithm (Missing, Switch or Discontinuation = Failure). Analysis was performed using a stratified analysis with CMH weights, adjusting for Baseline plasma HIV-1 RNA ( =<versus [vs]. >100,000 c/mL) and CD4+ cell count (=<350 cells/mm^3 or >350 cells/mm^3). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT population. Percentage values are rounded off.
Time Frame: Week 48
Population: as for outcome 40
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 248 | 247
Percentage of participants
  Age, <50 Years, n=212, 212: number analyzed (Participants) | 212 | 212
  Age, <50 Years, n=212, 212 | 80 | 71
  Age, >=50 Years, n=36, 35: number analyzed (Participants) | 36 | 35
  Age, >=50 Years, n=36, 35 | 92 | 74
  Race, White, n=115, 107: number analyzed (Participants) | 115 | 107
  Race, White, n=115, 107 | 86 | 80
  Race, Non-White, n=133,140: number analyzed (Participants) | 133 | 140
  Race, Non-White, n=133,140 | 78 | 64
  Race, African-American/African Heritage, n=102,108: number analyzed (Participants) | 102 | 108
  Race, African-American/African Heritage, n=102,108 | 74 | 67
  Non-African-American/African Heritage, n=146, 139: number analyzed (Participants) | 146 | 139
  Non-African-American/African Heritage, n=146, 139 | 88 | 75
  BPHR, <1000, n=5, 10: number analyzed (Participants) | 5 | 10
  BPHR, <1000, n=5, 10 | 60 | 80
  BPHR, 1000 to <10,000, n=66, 62: number analyzed (Participants) | 66 | 62
  BPHR, 1000 to <10,000, n=66, 62 | 83 | 77
  BPHR, 10,000 to <50,000, n=83, 81: number analyzed (Participants) | 83 | 81
  BPHR, 10,000 to <50,000, n=83, 81 | 84 | 74
  BPHR, 50,000 to <=100,000, n=25, 28: number analyzed (Participants) | 25 | 28
  BPHR, 50,000 to <=100,000, n=25, 28 | 80 | 64
  BPHR, >100,000, n=69, 66: number analyzed (Participants) | 69 | 66
  BPHR, >100,000, n=69, 66 | 80 | 64
  BCCC, <200, n=64, 49: number analyzed (Participants) | 64 | 49
  BCCC, <200, n=64, 49 | 81 | 69
  BCCC, >=200, n=184, 198: number analyzed (Participants) | 184 | 198
  BCCC, >=200, n=184, 198 | 82 | 72
  BCCC, <50, n=9, 15: number analyzed (Participants) | 9 | 15
  BCCC, <50, n=9, 15 | 67 | 60
  BCCC, 50 to <200, n=55, 34: number analyzed (Participants) | 55 | 34
  BCCC, 50 to <200, n=55, 34 | 84 | 74
  BCCC, 200 to <350, n=66, 74: number analyzed (Participants) | 66 | 74
  BCCC, 200 to <350, n=66, 74 | 89 | 73
  BCCC, 350 to <500, n=56, 65: number analyzed (Participants) | 56 | 65
  BCCC, 350 to <500, n=56, 65 | 79 | 74
  BCCC, >=500, n=62, 59: number analyzed (Participants) | 62 | 59
  BCCC, >=500, n=62, 59 | 77 | 68
  CDC category, A, n=210, 208: number analyzed (Participants) | 210 | 208
  CDC category, A, n=210, 208 | 81 | 71
  CDC category, B, n=27, 30: number analyzed (Participants) | 27 | 30
  CDC category, B, n=27, 30 | 81 | 77
  CDC category, C, n=11, 9: number analyzed (Participants) | 11 | 9
  CDC category, C, n=11, 9 | 91 | 56
  HIV-1 subtype: B vs Non-B, B, n=95, 111: number analyzed (Participants) | 95 | 111
  HIV-1 subtype: B vs Non-B, B, n=95, 111 | 80 | 69
  HIV-1 subtype: B vs Non-B, non-B, n=140, 131: number analyzed (Participants) | 140 | 131
  HIV-1 subtype: B vs Non-B, non-B, n=140, 131 | 84 | 73
  Argentina, n=24, 20: number analyzed (Participants) | 24 | 20
  Argentina, n=24, 20 | 92 | 80
  Canada, n=11, 9: number analyzed (Participants) | 11 | 9
  Canada, n=11, 9 | 91 | 89
  France, n=7, 8: number analyzed (Participants) | 7 | 8
  France, n=7, 8 | 100 | 75
  Italy, n=17, 11: number analyzed (Participants) | 17 | 11
  Italy, n=17, 11 | 88 | 64
  Mexico, n=6, 5: number analyzed (Participants) | 6 | 5
  Mexico, n=6, 5 | 100 | 60
  Portugal, n=4, 5: number analyzed (Participants) | 4 | 5
  Portugal, n=4, 5 | 75 | 60
  Puerto Rico, n=0, 2: number analyzed (Participants) | 0 | 2
  Puerto Rico, n=0, 2 |  | 100
  Russia, n=28, 22: number analyzed (Participants) | 28 | 22
  Russia, n=28, 22 | 89 | 82
  South Africa, n=33, 33: number analyzed (Participants) | 33 | 33
  South Africa, n=33, 33 | 67 | 76
  Spain, n=23, 31: number analyzed (Participants) | 23 | 31
  Spain, n=23, 31 | 70 | 77
  Thailand, n=19, 21: number analyzed (Participants) | 19 | 21
  Thailand, n=19, 21 | 95 | 52
  USA, n=62, 69: number analyzed (Participants) | 62 | 69
  USA, n=62, 69 | 74 | 67
  United Kingdom, n=14, 11: number analyzed (Participants) | 14 | 11
  United Kingdom, n=14, 11 | 93 | 64

43. Secondary Outcome: Number of Participants With Post-Baseline HIV-1 Disease Progression-Randomized Phase
Description: Number of participants with post-Baseline HIV-1disease progression were assessed during study period. The CDC Classification System for HIV Infection is the medical classification system used by the United States Centers for Disease Control and Prevention (CDC) to classify HIV disease and infection. The clinical categories of HIV infection are defined as follows: Category A: Mildly symptomatic, Category B: Moderately symptomatic, Category C: Severely symptomatic. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. Only those participants available at the specified time points were analyzed. Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT population.
Time Frame: Up to week 48
Population: ITT-E Population, only those participants who experienced a disease progression to CDC Class C or death were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase
Number analyzed (Participants) | 7 | 7
Participants
  CDC Class A to CDC Class C | 5 | 4
  CDC Class B to CDC Class C | 1 | 2
  CDC Class C to new CDC Class C | 0 | 0
  CDC Class A, B or C to Death | 1 | 1

44. Secondary Outcome: Number of Participants With Post-Baseline HIV-1 Disease Progression for DTG 50 mg/ABC 600 mg/3TC 300 mg QD (Randomized + Continuation Phase)
Description: as for outcome 43
Time Frame: Up to week 432
Population: ITT-E Population, only those participants who experienced a disease progression to CDC Class C or death were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- DTG 50 mg/ABC 600 mg/3TC 300 mg QD: Participants received fixed dose combination (FDC) of DTG/ABC/3TC 50 milligram (mg)/600 mg/300 mg tablet once daily orally for 48 weeks in the Randomization Phase. Participants who completed 48 weeks of treatment, continued to receive DTG/ABC/3TC in the Continuation Phase until it was either locally approved or commercial supplies were available.
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD
Number analyzed (Participants) | 9
Participants
  CDC Class A to CDC Class C | 6
  CDC Class B to CDC Class C | 1
  CDC Class C to new CDC Class C | 0
  CDC Class A, B or C to Death | 2

45. Secondary Outcome: Number of Participants With Treatment Emergent Resistances for DTG 50 mg/ABC 600 mg/3TC 300 mg QD (Randomized + Continuation Phase)
Description: Number of participants, who meet confirmed virologic withdrawal criteria, with treatment emergent genotypic resistance to integrase strand transfer inhibitor (INSTI), Non-nucleoside reverse transcriptase inhibitor (NNRTI), nucleoside reverse transcriptase inhibitor (NRTI), protease inhibitors (PI) will be summarized. The Baseline value was defined as the latest pre-dose assessment (Day 1) value. On-treatment Genotypic Resistance Population comprised of all participants in the ITTE population with available On-treatment genotypic resistance data at the time confirmed virologic withdrawal criterion was met.
Time Frame: Up to week 432
Population: On-treatment Genotypic Resistance Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD
Number analyzed (Participants) | 8
Participants
  INSTI; n= 6: number analyzed (Participants) | 6
  INSTI; n= 6 | 0
  NNRTI; n=8 | 1
  NRTI; n=8 | 1
  PI; n=8 | 0

46. Secondary Outcome: Number of Participants With Treatment Emergent Resistances for ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200mg QD (Randomized Phase)
Description: as for outcome 45
Time Frame: Up to week 48
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Groups:
- ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200mg QD-Randomized Phase: Participants received ATV 300 mg capsule, RTV 100 mg tablet, TDF/FTC FDC 300 mg/200 mg tablet once daily orally for 48 weeks during Randomized Phase
Arm/Group | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200mg QD-Randomized Phase
Number analyzed (Participants) | 4
Participants
  INSTI; n= 3: number analyzed (Participants) | 3
  INSTI; n= 3 | 1
  NNRTI; n=4 | 0
  NRTI; n=4 | 1
  PI; n=4 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs) and non-SAEs were collected up to Week 48 for Randomized Phase; from Weeks 48 to 432 for Continuation Phase
Description: All-Cause Mortality, SAEs and non-SAEs were reported for the Safety Population for the Randomized Phase, which comprised of all randomized participants who received at least one dose of study treatment. Safety-Continuation Population was used for the Continuation Phase which comprised of all participants in the DTG/ABC/3TC group who received at least 1 dose of study treatment after entering the Continuation Phase.
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase
All-Cause Mortality (participants affected / at risk) | 1/248 | 0/247 | 1/149
Serious Adverse Events (participants affected / at risk) | 12/248 | 20/247 | 13/149
Other Adverse Events (participants affected / at risk) | 138/248 | 164/247 | 30/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase (N=248) | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase (N=247) | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase (N=149)
Pneumonia (Infections and infestations) | 1 | 2 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 2
Acute hepatitis C (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Randomized Phase (N=248) | ATV 300 mg+RTV 100 mg+TDF 300 mg/FTC 200 mg QD-Randomized Phase (N=247) | DTG 50 mg/ABC 600 mg/3TC 300 mg QD-Continuation Phase (N=149)
Nausea (Gastrointestinal disorders) | 46 | 49 | 0
Diarrhoea (Gastrointestinal disorders) | 23 | 32 | 8
Dyspepsia (Gastrointestinal disorders) | 9 | 25 | 0
Vomiting (Gastrointestinal disorders) | 15 | 18 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 17 | 0
Upper respiratory tract infection (Infections and infestations) | 18 | 21 | 13
Nasopharyngitis (Infections and infestations) | 15 | 14 | 0
Urinary tract infection (Infections and infestations) | 13 | 17 | 9
Headache (Nervous system disorders) | 29 | 32 | 12
Dizziness (Nervous system disorders) | 13 | 15 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 26 | 0
Rash (Skin and subcutaneous tissue disorders) | 13 | 21 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 18 | 0
Jaundice (Hepatobiliary disorders) | 0 | 14 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 13 | 0
Fatigue (General disorders) | 8 | 15 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 18 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 8 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT01910402/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT01910402/SAP_001.pdf